CLINICAL TRIAL: NCT00006488
Title: Continuously Infused Intracerebral (IC) Recombinant-Methionyl Human Glial Cell Line-Derived Neurotrophic Factor (r-metHuGDNF) for the Treatment of Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00096-0968; M01RR000096 (NIH)
Record Dates: First submitted 2000-11-08; First posted 2000-11-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: recombinant-methionyl human glial cell line-derived neurotrophic factor

SUMMARY:
Parkinson's disease is characterized by loss of neurons that produce dopamine in a region of the brain called the substantia nigra. In the early stages of the disease, the disease responds to agents that replace dopamine such as levodopa. Patients with more advanced disease have wide fluctuations in their response to levodopa, exhibiting on and off periods. This is due to continued degeneration of neurons. Recombinant-methionyl human glial cell line-derived neurotrophic factor (r-metHuGDNF or GDNF) is a neurotrophic factor that promotes survival of dopaminergic neurons. This is a protein produced by recombinant technology that is almost identical to the naturally produced factor. Results of animal studies indicate that GDNF has the potential to benefit patients with advanced Parkinson's disease.

The purpose of this clinical trial is to determine whether GDNF works to relieve symptoms of advanced Parkinson's disease. The study will also test the delivery of GDNF using a catheter implanted into the putamen, the area of the brain associated with Parkinson's disease, and an infusion pump that is implanted under the skin in the abdomen or chest. GDNF will be placed into the pump and delivered through the catheter to the brain. The purposes of this study are to determine the potential benefits and side effects of GDNF. The performance and safety of the catheter/infusion pump system will also be assessed. The study will last for 6 months. Subjects will undergo neurological testing, computerized gait assessment and neurological imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced idiopathic Parkinson's disease treated with optimal doses of levodopa, dopamine agonist, catechol-o-methyl transferase (COMT) inhibitors, or selegiline for 2 months prior to implantation of the intracerebral catheter and pump.
* Must be able to undergo surgery required to implant the pump and catheter.
* Must be capable of informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, New York, New York, United States